CLINICAL TRIAL: NCT01655173
Title: Cognitive Behavioural Therapy and Recreational Activity for Adults With Autism Spectrum Disorders. A Randomized Controlled Trial.
Brief Title: Cognitive Behavioural Therapy (CBT) and Recreational Activity for Autism Spectrum Disorders (ASD)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Karolinska Institutet (Other)
Collaborators: Ministry of Health and Social Affairs, Sweden (Other Government)
Responsible Party: Principal Investigator, Susanne Bejerot, Associate professor, Karolinska Institutet
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Dnr 52-6104
Record Dates: First submitted 2012-07-25; First posted 2012-08-01 (Estimated); Last update posted 2020-10-22 (Actual); Status verified 2020-10

CONDITIONS: Asperger Syndrome; Autistic Disorder; Atypical Autism
Keywords: Asperger syndrome; Autistic disorder; Adult; Psychotherapy
MeSH Terms: conditions — Asperger Syndrome; Autistic Disorder | interventions — Cognitive Behavioral Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Cognitive behaviour therapy (Experimental): 36 weekly sessions (1 calendar year) of Cognitive behaviour therapy in a group setting.
  Interventions: Behavioral: Cognitive behaviour therapy
- Recreational activity intervention (Active Comparator): 36 sessions (1 calendar year) of a group intervention to enable social interaction and to break social isolation.
  Interventions: Behavioral: Recreational activity intervention

INTERVENTIONS:
Behavioral: Cognitive behaviour therapy — The CBT intervention consisted of five elements: (a) structure, (b) group setting, (c) psycho-education, (d) social training and (e) CBT.
  The participants were presented with the session plan for the whole year and given a binder in which they kept all materials. In addition, each session followed a strict agenda: (1) introduction and presentation of the agenda of the day, (2) resume of homework assignments from the previous session, (3) psycho-educative lecture and discussions on the session topic, (4) coffee break with buns or sandwiches, and social interaction, (5) relaxation or mindfulness exercise, (6) discussions and exercises on the session topic, (7) distribution of homework and (8) evaluation and end of session.
  Arms: Cognitive behaviour therapy
Behavioral: Recreational activity intervention — The therapists did not provide any deliberate interventions, such as psychoeducation, social training or CBT. Instead, the intervention relied on structure and group setting only. During the first session the participants were asked to write down group activities they would like to engage in. The therapists created a list of the suggested activities, such as visiting museums, board game playing, cooking, restaurant visits, boating, cinema and taking walks. The participants voted for the activity of the next session.
  Arms: Recreational activity intervention

SUMMARY:
The purpose of this study is to determine if adults with autism spectrum disorder and with normal intelligence improve from 36 sessions (1 calendar year) of group treatment with Cognitive Behavioural Therapy or recreational activity in groups with 6-8 participants.

DETAILED DESCRIPTION:
The purpose of this study was to compare two group interventions for psychiatric patients with Autism spectrum disorder and normal intelligence: Cognitive Behavioural Therapy developed to suit adults with Autism spectrum disorder, and recreational activity, enabling social interaction. The recreational activity intervention served as a low-impact option, easily organised within the community. It is not a placebo; rather it controls for the positive effects that come out of a structured social environment and group setting. The investigators hypothesized that both interventions would lead to improvement in quality of life, well-being and relief in psychiatric symptoms, with a greater effect in the Cognitive Behavioural Therapy intervention compared to recreational activity. A cumulative follow-up was made, within 5 1/2 years after the start of the treatments. Additional questions adapted to the patient group were added at this 5 1/2 year time point.

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of autism spectrum disorders
* Normal intelligence as assumed by mainstream schooling
* Acceptance of a group setting
* Being able to transport themselves to the clinic (with or without support)

Exclusion Criteria:

* Current substance abuse
* Current psychosis

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 68 (Actual)
Dates: Start 2005-08; Primary Completion 2011-09 (Actual); Study Completion 2011-09 (Actual)

PRIMARY OUTCOMES:
The Quality of Life Inventory (QOLI, Frisch et al. 1992) | Baseline, after 36 sessions (1 calendar year) and at a cumulative follow-up within 5 years after treatment termination
  Changes in the Quality of Life Inventory from baseline.
Sense of Coherence (SoC, Antonovsky 1993) | At baseline and after 36 sessions (1 calendar year)
  Self-rating scale, change from baseline
The ten-item Rosenberg Self Esteem Scale (RSES, Rosenberg 1962) | Before treatment (baseline) and after 36 sessions (1 calendar year)
  This was used to measure self esteem, change from baseline.
The patient versions of the Clinical Global Impression scale - Severity (patient CGI-S) | Before treatment and after 36 sessions (1 calendar year)
  Severity of impairment at baseline rated by the patient. Change from baseline.
Clinical Global Impression scale - Improvement (patient CGI-I) | Before treatment (at baseline) and at a cumulative follow-up within 5 years after treatment termination
  Patient rating on a seven-step Likert scale

SECONDARY OUTCOMES:
Autism Quotient (AQ, Baron-Cohen et al. 2001) | At baseline and after 36 sessions (1 calendar year)
  A 50-item screening instrument for measuring autistic traits. Change from baseline.
Adult ADHD Self-Report Scale (ASRS, Kessler et al. 2005) | At baseline and after 36 sessions (1 calendar year)
  This is for self rating scale for measuring inattention, hyperactivity and impulsivity.
Beck Depression Inventory (BDI, Beck et al. 1996) | At baseline and after 36 sessions (1 calendar year)
  This is a 20-item questionnaire to assess depression.
Symptom Checklist 90 (SCL-90, Derogatis & Cleary 1977) | At baseline and after 36 sessions (1 calendar year)
  This is a 90-item self rating questionnaire assessing the presence and severity of various psychiatric symptoms

OTHER OUTCOMES:
Drop-out | After 36 sessions (1 calendar year)
  How many sessions that each patient attended of the 36 sessions.

CONTACTS AND LOCATIONS:
Overall Officials: Susanne Bejerot, MD, PhD, Principal Investigator — Karolinska Institutet
Locations (1):
- Northern Stockholm psychiatry, St. Göran hospital, Stockholm, Sweden

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Result] Hesselmark E, Plenty S, Bejerot S. Group cognitive behavioural therapy and group recreational activity for adults with autism spectrum disorders: a preliminary randomized controlled trial. Autism. 2014 Aug;18(6):672-83. doi: 10.1177/1362361313493681. Epub 2013 Oct 2. PMID 24089423
- See also: PMID: 24089423 — https://www-ncbi-nlm-nih-gov.proxy.kib.ki.se/pmc/articles/PMC4230566/